CLINICAL TRIAL: NCT04438187
Title: Trial of Antimicrobial Restraint in Presumed Pneumonia
Acronym: TARPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Western Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 145059
Record Dates: First submitted 2020-06-08; First posted 2020-06-18 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthcare-Associated Pneumonia; Sepsis
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Sepsis

STUDY DESIGN:
Intervention Model Description: This will be a pragmatic, before-and-after, cluster-randomized, protocol crossover study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aggressive Arm (Other): If an intubated patient is suspected of having an ICU-acquired HAP/VAP during the aggressive period, antimicrobials should be initiated immediately after quantitative or semi-quantitative endobronchial cultures are sent regardless of clinical status. This will include patients who, as determined by the attending intensivist, are in sepsis or septic shock. If, after 72 hours, cultures and other clinical data do not point to a pneumonia, the antimicrobials should be stopped in the absence of another source of infection.
  Interventions: Other: antimicrobial initiation
- Conservative Arm (Other): If a patient is suspected of having an ICU-acquired HAP/VAP during the conservative period, quantitative or semi-quantitative endobronchial cultures should be sent. If the patient is in septic shock persistent hypotension requiring vasoactive medications to maintain mean arterial pressure (MAP) ≥65 mm HG or persistent lactic acidosis (>2 mmol/L) despite adequate resuscitation) antimicrobials will be initiated immediately. If the patient has new onset organ dysfunction that is presumed to be due to infection (sepsis) then antimicrobials will be initiated at the discretion of the attending intensivist. In the absence of septic shock or sepsis (intensivist discretion), antimicrobials will not be initiated unless objective evidence of pneumonia is present or another documented source of infection is identified mandating treatment with antimicrobials.
  Interventions: Other: antimicrobial initiation

INTERVENTIONS:
Other: antimicrobial initiation — antimicrobial initiation based on protocol assignment.

SUMMARY:
The objective of this cluster-randomized crossover study is to determine the effect of delaying antimicrobial initiation until objective microbiologic data is obtained in patients with presumed ICU-acquired pneumonia without septic shock.

DETAILED DESCRIPTION:
This study will involve 8 centers is to determine the effect of delaying antimicrobial initiation until objective microbiologic data is obtained in patients with presumed ICU-acquired pneumonia without septic shock. The study team will compare two sequential 4-month periods in each unit, one 'aggressive' antimicrobial initiation period and one 'conservative' antimicrobial initiation period.

This study will serve the following specific aims:

Specific Aim 1: To determine feasibility of a larger multicenter study of the same design as well as assess protocol adherence across multiple centers.

Specific Aim 2: Prospectively determine the all-cause, in-hospital mortality for all patients with suspected pneumonia who were treated under either an aggressive or conservative antimicrobial initiation protocol.

Specific Aim 3: Prospectively determine antimicrobial initiation rates, total days of antimicrobial administration, hospital and ICU length of stay, and ventilator-free alive days for patients treated under each protocol.

Specific Aim 4: To survey physicians that participated in the study to assess their feelings about the study including level of comfort starting antimicrobials aggressively, level of comfort withholding antimicrobials until definitive evidence of infection, perceived protocol adherence, perceived importance of the study, and willingness to participate in other studies of its kind (to be performed after closure of the clinical portion of the study).

ELIGIBILITY:
Inclusion Criteria:

* Intubated patients admitted to a surgical or trauma intensive care unit that have had an appropriate quantitative or semi-quantitative endobronchial sputum culture sent ≥48 hours into their ICU admission
* Primary pathology managed by surgical specialty
* Age ≥18 years.

Exclusion Criteria:

* Non-intubated patients.
* Intubated patients with concern for active infection that is not suspected to be pneumonia (i.e. intra-abdominal infection, skin and soft tissue infection, urinary tract infection, etc.)
* Primary disease not surgical or traumatic in nature
* Primary diagnosis of burns
* Incarcerated status
* Pregnant status or delivery during this hospitalization.
* On active immunosuppressive medications (or taking as a home medication prior to arrival)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
protocol adherence | by time of culture finalization or 1 week
  as a pilot study the primary outcome will be protocol adherence as defined by using the criteria below:
  Aggressive Protocol:
  * Failure to send appropriate culture before initiation of antimicrobials in the absence of septic shock
  * Failure to stop antimicrobials in the absence of pneumonia or other documented infection after 72 hours.
  Conservative Protocol:
  * Failure to send appropriate culture
  * Initiation of antimicrobials (in the absence of septic shock, new onset or worsening organ dysfunction, or other indicated source of infection) without any objective evidence of pneumonia.
  * Failure to initiate antimicrobials in the setting of objective evidence of pneumonia.
  * Failure to stop antimicrobials in the absence of other documented infection if final cultures return as negative.

SECONDARY OUTCOMES:
In-hospital mortality | until hospital discharge or 1 year
  All-cause, by treatment protocol assignment (intent-to-treat), ICU mortality, pneumonia-related
Days of antimicrobials administered | until hospital discharge or 1 year
  includes empiric, therapeutic, prophylactic, and perioperative antimicrobials
Ventilator-free alive days | until hospital discharge or 1 year
ICU length of stay | Until discharge from ICU or 1 year
Hospital length of stay | until hospital discharge or 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Guidry, Principal Investigator — KU Medical Center
Locations (1):
- KU Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
aggregated study results

REFERENCES:
- [Background] Hranjec T, Rosenberger LH, Swenson B, Metzger R, Flohr TR, Politano AD, Riccio LM, Popovsky KA, Sawyer RG. Aggressive versus conservative initiation of antimicrobial treatment in critically ill surgical patients with suspected intensive-care-unit-acquired infection: a quasi-experimental, before and after observational cohort study. Lancet Infect Dis. 2012 Oct;12(10):774-80. doi: 10.1016/S1473-3099(12)70151-2. Epub 2012 Aug 28. PMID 22951600
- [Background] Barbier F, Andremont A, Wolff M, Bouadma L. Hospital-acquired pneumonia and ventilator-associated pneumonia: recent advances in epidemiology and management. Curr Opin Pulm Med. 2013 May;19(3):216-28. doi: 10.1097/MCP.0b013e32835f27be. PMID 23524477
- [Background] Torres A, Niederman MS, Chastre J, Ewig S, Fernandez-Vandellos P, Hanberger H, Kollef M, Li Bassi G, Luna CM, Martin-Loeches I, Paiva JA, Read RC, Rigau D, Timsit JF, Welte T, Wunderink R. International ERS/ESICM/ESCMID/ALAT guidelines for the management of hospital-acquired pneumonia and ventilator-associated pneumonia: Guidelines for the management of hospital-acquired pneumonia (HAP)/ventilator-associated pneumonia (VAP) of the European Respiratory Society (ERS), European Society of Intensive Care Medicine (ESICM), European Society of Clinical Microbiology and Infectious Diseases (ESCMID) and Asociacion Latinoamericana del Torax (ALAT). Eur Respir J. 2017 Sep 10;50(3):1700582. doi: 10.1183/13993003.00582-2017. Print 2017 Sep. PMID 28890434
- [Background] Leonard KL, Borst GM, Davies SW, Coogan M, Waibel BH, Poulin NR, Bard MR, Goettler CE, Rinehart SM, Toschlog EA. Ventilator-Associated Pneumonia in Trauma Patients: Different Criteria, Different Rates. Surg Infect (Larchmt). 2016 Jun;17(3):363-8. doi: 10.1089/sur.2014.076. Epub 2016 Mar 3. PMID 26938612
- [Background] Krebs ED, Hassinger TE, Guidry CA, Berry PS, Elwood NR, Sawyer RG. Non-utility of sepsis scores for identifying infection in surgical intensive care unit patients. Am J Surg. 2019 Aug;218(2):243-247. doi: 10.1016/j.amjsurg.2018.11.044. Epub 2018 Dec 8. PMID 30553458
- [Background] Eguia E, Cobb AN, Baker MS, Joyce C, Gilbert E, Gonzalez R, Afshar M, Churpek MM. Risk factors for infection and evaluation of Sepsis-3 in patients with trauma. Am J Surg. 2019 Nov;218(5):851-857. doi: 10.1016/j.amjsurg.2019.03.005. Epub 2019 Mar 8. PMID 30885453
- [Background] Anand V, Zhang Z, Kadri SS, Klompas M, Rhee C; CDC Prevention Epicenters Program. Epidemiology of Quick Sequential Organ Failure Assessment Criteria in Undifferentiated Patients and Association With Suspected Infection and Sepsis. Chest. 2019 Aug;156(2):289-297. doi: 10.1016/j.chest.2019.03.032. Epub 2019 Apr 9. PMID 30978329
- [Background] Piriyapatsom A, Lin H, Pirrone M, De Pascale G, Corona De Lapuerta J, Bittner EA, Schmidt UH, De Moya M, Berra L. Evaluation of the Infection-Related Ventilator-Associated Events Algorithm for Ventilator-Associated Pneumonia Surveillance in a Trauma Population. Respir Care. 2016 Mar;61(3):269-76. doi: 10.4187/respcare.04280. Epub 2015 Nov 10. PMID 26556896
- [Background] Pieracci FM, Rodil M, Haenel J, Stovall RT, Johnson JL, Burlew CC, Jurkovich GJ, Moore EE. Screening for Ventilator-Associated Pneumonia in the Surgical Intensive Care Unit: A Single-Institution Analysis of 1,013 Lower Respiratory Tract Cultures. Surg Infect (Larchmt). 2015 Aug;16(4):368-74. doi: 10.1089/sur.2014.086. Epub 2015 May 28. PMID 26207397
- [Background] Carraro E, Cook C, Evans D, Stawicki S, Postoev A, Olcese V, Phillips G, Eiferman D. Lack of added predictive value of portable chest radiography in diagnosing ventilator-associated pulmonary infection. Surg Infect (Larchmt). 2014 Dec;15(6):739-44. doi: 10.1089/sur.2013.239. PMID 25314257
- [Background] Croce MA, Swanson JM, Magnotti LJ, Claridge JA, Weinberg JA, Wood GC, Boucher BA, Fabian TC. The futility of the clinical pulmonary infection score in trauma patients. J Trauma. 2006 Mar;60(3):523-7; discussion 527-8. doi: 10.1097/01.ta.0000204033.78125.1b. PMID 16531849
- [Background] Quick JA, Breite MD, Barnes SL. Inadequacy of Algorithmic Ventilator-Associated Pneumonia Diagnosis in Acute Care Surgery. Am Surg. 2018 Feb 1;84(2):300-304. PMID 29580362
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Background] Dellinger RP, Carlet JM, Masur H, Gerlach H, Calandra T, Cohen J, Gea-Banacloche J, Keh D, Marshall JC, Parker MM, Ramsay G, Zimmerman JL, Vincent JL, Levy MM; Surviving Sepsis Campaign Management Guidelines Committee. Surviving Sepsis Campaign guidelines for management of severe sepsis and septic shock. Crit Care Med. 2004 Mar;32(3):858-73. doi: 10.1097/01.ccm.0000117317.18092.e4. PMID 15090974
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Crit Care Med. 2017 Mar;45(3):486-552. doi: 10.1097/CCM.0000000000002255. PMID 28098591
- [Background] Barie PS, Hydo LJ, Shou J, Larone DH, Eachempati SR. Influence of antibiotic therapy on mortality of critical surgical illness caused or complicated by infection. Surg Infect (Larchmt). 2005 Spring;6(1):41-54. doi: 10.1089/sur.2005.6.41. PMID 15865550
- [Background] Kumar A, Roberts D, Wood KE, Light B, Parrillo JE, Sharma S, Suppes R, Feinstein D, Zanotti S, Taiberg L, Gurka D, Kumar A, Cheang M. Duration of hypotension before initiation of effective antimicrobial therapy is the critical determinant of survival in human septic shock. Crit Care Med. 2006 Jun;34(6):1589-96. doi: 10.1097/01.CCM.0000217961.75225.E9. PMID 16625125
- [Background] Barochia AV, Cui X, Vitberg D, Suffredini AF, O'Grady NP, Banks SM, Minneci P, Kern SJ, Danner RL, Natanson C, Eichacker PQ. Bundled care for septic shock: an analysis of clinical trials. Crit Care Med. 2010 Feb;38(2):668-78. doi: 10.1097/CCM.0b013e3181cb0ddf. PMID 20029343
- [Background] Gaieski DF, Mikkelsen ME, Band RA, Pines JM, Massone R, Furia FF, Shofer FS, Goyal M. Impact of time to antibiotics on survival in patients with severe sepsis or septic shock in whom early goal-directed therapy was initiated in the emergency department. Crit Care Med. 2010 Apr;38(4):1045-53. doi: 10.1097/CCM.0b013e3181cc4824. PMID 20048677
- [Background] Ferrer R, Martin-Loeches I, Phillips G, Osborn TM, Townsend S, Dellinger RP, Artigas A, Schorr C, Levy MM. Empiric antibiotic treatment reduces mortality in severe sepsis and septic shock from the first hour: results from a guideline-based performance improvement program. Crit Care Med. 2014 Aug;42(8):1749-55. doi: 10.1097/CCM.0000000000000330. PMID 24717459
- [Background] Loftus TJ, Brakenridge SC, Moore FA, Lemon SJ, Nguyen LL, Voils SA, Jordan JR, Croft CA, Smith RS, Efron PA, Mohr AM. Intubated Trauma Patients Receiving Prolonged Antibiotics for Pneumonia despite Negative Cultures: Predictors and Outcomes. Surg Infect (Larchmt). 2016 Dec;17(6):766-772. doi: 10.1089/sur.2016.108. Epub 2016 Sep 16. PMID 27635693
- [Background] Klompas M, Calandra T, Singer M. Antibiotics for Sepsis-Finding the Equilibrium. JAMA. 2018 Oct 9;320(14):1433-1434. doi: 10.1001/jama.2018.12179. No abstract available. PMID 30242350
- [Background] Mi MY, Klompas M, Evans L. Early Administration of Antibiotics for Suspected Sepsis. N Engl J Med. 2019 Feb 7;380(6):593-596. doi: 10.1056/NEJMclde1809210. No abstract available. PMID 30726686
- [Background] Prescott HC, Iwashyna TJ. Improving Sepsis Treatment by Embracing Diagnostic Uncertainty. Ann Am Thorac Soc. 2019 Apr;16(4):426-429. doi: 10.1513/AnnalsATS.201809-646PS. No abstract available. PMID 30883190
- [Background] Alam N, Oskam E, Stassen PM, Exter PV, van de Ven PM, Haak HR, Holleman F, Zanten AV, Leeuwen-Nguyen HV, Bon V, Duineveld BAM, Nannan Panday RS, Kramer MHH, Nanayakkara PWB; PHANTASi Trial Investigators and the ORCA (Onderzoeks Consortium Acute Geneeskunde) Research Consortium the Netherlands. Prehospital antibiotics in the ambulance for sepsis: a multicentre, open label, randomised trial. Lancet Respir Med. 2018 Jan;6(1):40-50. doi: 10.1016/S2213-2600(17)30469-1. Epub 2017 Nov 28. PMID 29196046
- [Background] Bloos F, Thomas-Ruddel D, Ruddel H, Engel C, Schwarzkopf D, Marshall JC, Harbarth S, Simon P, Riessen R, Keh D, Dey K, Weiss M, Toussaint S, Schadler D, Weyland A, Ragaller M, Schwarzkopf K, Eiche J, Kuhnle G, Hoyer H, Hartog C, Kaisers U, Reinhart K; MEDUSA Study Group. Impact of compliance with infection management guidelines on outcome in patients with severe sepsis: a prospective observational multi-center study. Crit Care. 2014 Mar 3;18(2):R42. doi: 10.1186/cc13755. PMID 24589043
- [Background] Abe T, Ogura H, Shiraishi A, Kushimoto S, Saitoh D, Fujishima S, Mayumi T, Shiino Y, Nakada TA, Tarui T, Hifumi T, Otomo Y, Okamoto K, Umemura Y, Kotani J, Sakamoto Y, Sasaki J, Shiraishi SI, Takuma K, Tsuruta R, Hagiwara A, Yamakawa K, Masuno T, Takeyama N, Yamashita N, Ikeda H, Ueyama M, Fujimi S, Gando S; JAAM FORECAST group. Characteristics, management, and in-hospital mortality among patients with severe sepsis in intensive care units in Japan: the FORECAST study. Crit Care. 2018 Nov 22;22(1):322. doi: 10.1186/s13054-018-2186-7. PMID 30466493
- [Background] de Groot B, Ansems A, Gerling DH, Rijpsma D, van Amstel P, Linzel D, Kostense PJ, Jonker M, de Jonge E. The association between time to antibiotics and relevant clinical outcomes in emergency department patients with various stages of sepsis: a prospective multi-center study. Crit Care. 2015 Apr 29;19(1):194. doi: 10.1186/s13054-015-0936-3. PMID 25925412
- [Background] Kaasch AJ, Rieg S, Kuetscher J, Brodt HR, Widmann T, Herrmann M, Meyer C, Welte T, Kern P, Haars U, Reuter S, Hubner I, Strauss R, Sinha B, Brunkhorst FM, Hellmich M, Fatkenheuer G, Kern WV, Seifert H; preSABATO study group. Delay in the administration of appropriate antimicrobial therapy in Staphylococcus aureus bloodstream infection: a prospective multicenter hospital-based cohort study. Infection. 2013 Oct;41(5):979-85. doi: 10.1007/s15010-013-0428-9. Epub 2013 Mar 29. PMID 23539143
- [Derived] Guidry CA, Beyene RT, Watson CM, Sawyer RG, Chollet-Hinton L, Simpson SQ, Atchison L, Derickson M, Cooper LC, Pennington GP 2nd, VandenBerg S, Halimeh BN, O'Dell JC. Trial of antibiotic restraint in presumed pneumonia: A Surgical Infection Society multicenter pilot. J Trauma Acute Care Surg. 2023 Feb 1;94(2):232-240. doi: 10.1097/TA.0000000000003839. Epub 2022 Nov 18. PMID 36534474
- See also: Trial of antibiotic restraint in presumed pneumonia: A Surgical Infection Society multicenter pilot — http://pubmed.ncbi.nlm.nih.gov/36534474/